CLINICAL TRIAL: NCT05034588
Title: Multiparametric Cardiac MRI for the Detection and Quantification of Myocardial Injury Following Acute Kidney Injury (Cardiorenal Syndrome Type 3)
Brief Title: Cardiac MRI for the Detection of Myocardial Injury Following Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Principal Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 519/20
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Acute Kidney Injury; Cardio-Renal Syndrome; Cardiomyopathies
Keywords: Cardiac MRI
MeSH Terms: conditions — Acute Kidney Injury; Cardio-Renal Syndrome; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensiv care patients after acute kidney injury: Patients with condition after intensive care stay and acute kidney injury and subsequent convalescence (without preexisting underlying cardiac disease or other disease with potential cardiac involvement).
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan
- Intensiv care patients without kidney injury: Patients with condition after intensive care stay and subsequent convalescence (without kidney injury and preexisting underlying cardiac disease or other disease with potential cardiac involvement).
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance scan — Multiparametric cardiac magnetic resonance, including functional and structural parameter

SUMMARY:
The aim of this clinical prospective study is to assess structural and functional myocardial changes in patients after acute kidney injury (Cardiorenal syndrome type 3) and intensive care stay by multiparametric cardiac MRI.

DETAILED DESCRIPTION:
The aim of the study is to demonstrate any differences in myocardial structure and function using multiparametric cardiac MRI in patients after acute kidney injury (Cardiorenal syndrome type 3) and intensive care stay and subsequent convalescence compared to a control group with intensive care stay but without kidney injury. Furthermore, the correlation between clinical disease severity and cardiac involvement will be investigated.

ELIGIBILITY:
Inclusion criteria:

1. acute kidney injury and convalescence (GFR > 45 ml/min/1.73m²).
2. patients who are 18 years of age or older

Exclusion criteria:

1. underlying cardiac disease, e.g. known myocardial infarction, previous myocarditis, congenital heart disease, cardiomyopathies of other causes
2. known underlying disease wit potential cardiac involvement, e.g. storage disease (e.g. hemochromatosis, Fabry disease), inflammatory (e.g. sarcoidosis), endocrinological (e.g. diabetes mellitus, hyper-/hypothyroidism), autoimmune (e.g. systemic lupus erythematosus, dermatomyositis, rheumatoid arthritis), therapeutic (chemotherapy).
3. patients with persistent renal failure and GFR < 45 ml/min/1.73m²
4. allergy to contrast media
5. patients who are using a intrauterinpessare for contraception
6. pregnant and breastfeeding women
7. patients with contraindications for MRI due to implants

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with convalescence after acute renal failure who were/are treated in the Department of Anesthesiology and Intensive Care Medicine of the University Hospital Bonn are included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial T1 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T1 relaxation times will be obtained to asses acute myocardial injury and fibrosis. T1 maps will be analyzed using a segmental approach by region of interest analysis. T1 relaxation times are given in [ms].

SECONDARY OUTCOMES:
Myocardial T2 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T2 relaxation times will be obtained to asses myocardial edema. T2 maps will be analyzed using a segmental approach by region of interest analysis. T2 relaxation times are given in [ms].
Myocardial ECV | Measurement will be performed within 2 weeks after MRI scan.
  Myocardial extracellular volume will be obtained to asses extracellular space/myocardial fibrosis. ECV values will be calculated using a segmental approach by region of interest analysis of native and contrast-enhanced T1 relaxation maps. ECV values are given in [%].
Myocardial strain | Measurement will be performed within 2 weeks after MRI scan.
  Cardiac magnetic resonance feature-tracking will be used to asses left ventricular longitudinal, circumferential and radial strain.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Department of Anesthesiology and Intensive Care Medicine, Bonn, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isaak A, Pomareda I, Mesropyan N, Kravchenko D, Endler C, Bischoff L, Pieper CC, Kuetting D, Attenberger U, Zimmer S, Putensen C, Schewe JC, Kreyer S, Luetkens JA. Cardiovascular Magnetic Resonance in Survivors of Critical Illness: Cardiac Abnormalities Are Associated With Acute Kidney Injury. J Am Heart Assoc. 2023 May 2;12(9):e029492. doi: 10.1161/JAHA.123.029492. Epub 2023 Apr 29. PMID 37119085